CLINICAL TRIAL: NCT05765929
Title: Use of Weightbearing Radiographs to Determine Treatment of bi- and Trimalleolar Ankle Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47891
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-11

CONDITIONS: Ankle Fracture, Bimalleolar; Ankle Fracture, Trimalleolar
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-operative treatment (Experimental): Non-operative treatment based on weightbearing radiographs
  Interventions: Other: Non-operative treatment

INTERVENTIONS:
Other: Non-operative treatment — Patients will be treated with a walker-orthosis for 6 weeks. Weightbearing as tolerated

SUMMARY:
The aim of this study is to evaluate the outcomes after non-operative treatment of weightbearing stable bi-and trimalleolar ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

* -With bi- and trimalleolar ankle fractures with less than 7 mm medial clear space on non-weightbearing radiographs that are deemed stable by weightbearing radiographs.
* With type B medial malleolus fractures between the tip and the plafond and type C medial malleolus fractures at the level of the plafond (Herscovici classification). (6)
* With fractures in the distal 1/3 of fibula (not-Maisonneuve)
* Enabling stability evaluation within 14 days after injury
* 18-75 years of age
* with pre-injury walking ability without aids

Exclusion Criteria:

* - With primary unstable ankle fractures, > 7mm medial clear space on primary radiographs
* With fracture reduction prior to initial radiographic evaluation, open fracture, fractures resulting from high-energy trauma or multi trauma and pathological fracture
* With type A medial malleolus avulsion fractures < 5mm (at the tip of the malleolus), that are not suitable for surgical intervention.
* With Herscovici type D fractures, involving Lauge-Hansen SA2 fractures (supracollicular fracture - vertical, oblique or transverse direction of the plafond)
* With displaced posterior malleolus fractures that needs fixation in the judgement of the attending surgeon
* With neuropathies and symptomatic joint diseases such as Rheumatoid Arthritis
* That are assumed not compliant (such as drug abuse, cognitive- and/or psychiatric disorders)
* With previous history ipsilateral ankle fracture
* With previous history ipsilateral major ankle-/foot surgery
* Who live outside the hospital catchment areas not available to follow up
* With insufficient Norwegian or English language skills
* Non-compliant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Olerud Molander Score (OMAS) to measure a change over time | 6 week, 12 weeks, 1year, 2 years
  Condition specific, patient reported measure of ankle-fracture symptoms

SECONDARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOxFQ) | 6 week, 12 weeks, 1year, 2 years
  Patients reported outcomes
Range of Motion measured by a goniometer (ad modum Lindsjo) | 6 week, 12 weeks, 1year, 2 years
  dorsiflexion and plantarflexion
Numeric Rating Scale (NRS) | 6 week, 12 weeks, 1year, 2 years
  Ankle pain in rest, at night and in daily activities, a 11-point numeric scale ranging from 0-10
Euroqol questionnaire (EQ- 5D) | 6 week, 12 weeks, 1year, 2 years
  Health related quality of life
Registrations of complications/adverse events | 0-2 years
  Registration of loss of congruence, delayed union, non-union, thromboembolic events
Posttraumatic osteoarthritis (OA) | 2 years and 5 years
  CT-scan (Kellgren-Lawrence classification)

CONTACTS AND LOCATIONS:
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No